CLINICAL TRIAL: NCT02677194
Title: Stimulation of Cutaneous Healing Processes With LED: a Controlled Comparative Study to Identify Optimal Settings
Brief Title: HeaLED: Pilot Study of Skin Healing Under LED Exposure
Acronym: HeaLed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-AOI-12
Record Dates: First submitted 2016-01-28; First posted 2016-02-09 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exposition LED (Experimental): The patient is his own witness. This is a randomization for the allocation of treatments (LED parameters) on 6 mini-zones of 1,5x1,5 cm at the level of forearm. Dermabrasion by fractional laser CO2 ablative, evaluation of the pain on every zone by VAS post-act : exposition to LED 590nm (4 or 12sec) or 630nm(4min30 or 15 min) or 830 nm (6 or 12 min).
  Interventions: Device: LED
- Control (Other): Device without any LED exposition : This is a randomization for the allocation of treatments (LED parameters) on 6 mini-zones of 1,5x1,5 cm at the level of forearm or control (1 mini-zone)
  Interventions: Other: Control device

INTERVENTIONS:
Device: LED — There are 7 mini-zones of 1,5x1,5 cm at the level of forearm, one of them is allocated to control ( only laser). Dermabrasion by fractional laser CO2 ablative, evaluation of the pain on every zone by VAS post-act. Exposition to LED (630nm, 830nm and 590 nm). Water loss measure and colorimetry before and after laser and after the exposition to LED. Clinical evaluation of local tolerance post-laser and post-LED + standardized photographs.
  Arms: Exposition LED
Other: Control device — Device without any LED exposition
  Arms: Control

SUMMARY:
The aim of this study is to assess cutaneous healing process under LED exposition on 10 healthy subjects pre-treated with fractional CO2 laser on mini-zones on forearms.

DETAILED DESCRIPTION:
Cutaneous healing is a physiological process that occurs in many occasions: posttraumatic, post-burn, but also in postsurgery or aesthetic interventions. Most often, topical products are used to create a favorable environment for wound healing.

LED (Light Emitting Diode) are light emitting diodes which produce monochromatic or non-coherent polychromatic radiation when an electric current passes through them. Some LED emitting wavelengths in the visible or near infrared have been reported to promote wound healing. In the literature, in vitro studies showed stimulation of fibroblast and keratinocyte proliferation under the effect of irradiation by the LED. Animal studies have also shown that some LED treatments were able to stimulate healing and angiogenesis. Despite existence of strong data in in vitro and animal studies, the clinical data in humans regarding wound healing are still very poor. Thus, it is still not clear whether the LEDs have a real interest in skin healing, and if so, what are the wavelengths and optimal parameters. Despite this, the LEDs are used widely, unfortunately without a clear demonstration of their effectiveness and without any determination of optimal parameters of treatments that could guide clinicians.

The main objective of the study is to evaluate the efficacy at day 3 of different parameters of LED to enhance wound healing after dermabrasion with CO2 fractional laser on mini-zones on 10 healthy volunteers.

Design of the study:

* screening visit (day-7 to day-21): information of the patient, verification of inclusion criteria , preselection of 7 mini-zones, collection of the informed consent. Clinical examination, vital signs. Pregnancy test for women old enough to procreate.
* V1 (inclusion): clinical examination, vital signs, new pregnancy test for the women old enough to procreate, randomization for the allocation of treatments (LED parameters) on 7 mini-zones of 1,5x1,5 cm at the level of forearm, one of them is allocated to control ( only laser). Dermabrasion by fractional laser CO2 ablative, evaluation of the pain on every zone by VAS post-act. Exposition to LED (630nm, 830nm and 590 nm). Water loss measure and colorimetry before and after laser and after the exposition to LED. Clinical evaluation of local tolerance post-laser and post-LED + standardized photographs. Application of a healing cream twice a day on area treated until healing.
* V2 (24 hours): evaluation local tolerance, photos, colorimetry, waterloss measure before the session LED.
* V3 (48 hours): evaluation local tolerance, photos, colorimetry, waterloss measure before the session LED
* V4 (72 hours): clinical exam, clinical local tolerance evaluation and healing, waterloss measure, colorimetry and standardized photos
* V5 ( J7): evaluation local tolerance, colorimetry and waterloss measures, standardized photos . V6 (J21+/-3 days): clinical exam, clinical local tolerance evaluation and healing, waterloss measure, colorimetry and standardized photos. Final visit of the study

ELIGIBILITY:
Inclusion Criteria:

* • Male or female aged 18 years or more

  * Phototype I to III
  * No allergy to topical anesthesia
  * Healthy subject with no medical history of dermatological or systemic disease
  * Normal homogeneous skin on forearms without excessive hair growth
  * No medical history of keloïds or hypertrophic scar
  * No history of post-inflammatory hyperpigmentation
  * No congenital methemoglobinemia or porphyria
  * No oral retinoids treatment in the 6 previous months before starting the study
  * No Topical or systemic corticosteroids or immunosuppressive or photosensitive drugs in the previous month
  * No medical issue that could interfere with the results of the study according to investigator opinion

Exclusion Criteria:

* • Subject within exclusion period according to the volunteer national file

  * Childbearing or breastfeeding women
  * Use of topical cosmetics or drugs in the 48 previous hour before inclusion
  * Antalgic treatment in the 24 previous hour before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Effect of LED treatement | at day 3
  The effect of LED treatment on skin healing will be estimated by measure on colorimetry (day 3 versus day 0)

SECONDARY OUTCOMES:
Waterloss measure | at day 3
  Compare waterloss measure at day 3 (V4) between different LED zones versus control zone by vaporimètre
Tolerance | at day 3 (V4)
  Describe LED effect on laser tolerance by scale EVA

CONTACTS AND LOCATIONS:
Overall Officials: Passeron Thierry, PhD, Principal Investigator — Centre Hospitalier Universitaire de Nice

IPD SHARING:
Plan to Share IPD: No